CLINICAL TRIAL: NCT00080873
Title: A Randomized Double Blind Placebo Controlled Clinical Trial to Assess the Efficacy of Traumeel® S (IND#66649) for the Prevention and Treatment of Mucositis in Children Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Traumeel® S in Preventing and Treating Mucositis in Young Patients Undergoing Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ACCL0331; CDR0000356179 (Other: Clinical Trials.gov); COG-ACCL0331 (Other: Children's Oncology Group); NCT00228800 (obsolete NCT alias)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2014-02

CONDITIONS: Kidney Cancer; Leukemia; Lymphoma; Neuroblastoma; Oral Complications; Sarcoma
Keywords: oral complications; disseminated neuroblastoma; previously treated childhood rhabdomyosarcoma; recurrent Wilms tumor and other childhood kidney tumors; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood rhabdomyosarcoma; recurrent childhood small noncleaved cell lymphoma; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; juvenile myelomonocytic leukemia; recurrent neuroblastoma
MeSH Terms: conditions — Kidney Neoplasms; Leukemia; Lymphoma; Neuroblastoma; Sarcoma; Wilms Tumor; Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Leukemia, Myelomonocytic, Juvenile | interventions — Traumeel S

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Receive Traumeel S (Experimental)
  Interventions: Drug: Traumeel S
- Receive placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Traumeel S
  Arms: Receive Traumeel S
Other: Placebo
  Arms: Receive placebo

SUMMARY:
RATIONALE: Traumeel® S (a mouth rinse) may be effective in preventing or decreasing the severity of oral mucositis caused by chemotherapy in young patients who are undergoing stem cell transplantation.

PURPOSE: This randomized clinical trial is studying how well Traumeel® S works in preventing or treating mucositis in young patients who are receiving chemotherapy with or without total-body irradiation before undergoing stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of Traumeel® S vs placebo in reducing the severity and duration of chemotherapy-induced (with or without total body irradiation) mucositis in pediatric patients undergoing hematopoietic stem cell transplantation.
* Determine the safety of this drug in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to treatment with total body irradiation during conditioning chemotherapy (yes vs no), type of transplantation (autologous vs allogeneic), and participating institution (COG vs foreign). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral Traumeel® S mouth rinse 5 times daily beginning on day -1 before transplantation.
* Arm II: Patients receive oral placebo mouth rinse 5 times daily beginning on day -1 before transplantation.

In both arms, treatment continues until day 20 post-transplantation OR until mucositis resolves to Walsh score ≤ 1 for 2 consecutive days.

Patients are followed until day 100 post-transplantation.

PROJECTED ACCRUAL: A total of 180 patients (90 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Planned treatment with allogeneic or autologous hematopoietic stem cell transplantation

  * Conditioning chemotherapy regimen for transplantation must be myeloablative
  * Source of stem cells from any of the following:

    * Bone marrow
    * Placental cord
    * Cytokine-mobilized peripheral blood
* Availability of 1 of the following donor types:

  * HLA-matched sibling or parent
  * Related donor mismatched for a single HLA locus (class I or II)
  * Unrelated marrow or peripheral blood stem cell donor
  * Unrelated umbilical cord blood HLA-matched or mismatched (class I) donor

PATIENT CHARACTERISTICS:

Age

* 3 to 25

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No known allergy to Echinacea
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent oral vancomycin paste
* No concurrent oral glutamine supplementation
* No other mouth care or oral medications within 30 minutes after administration of study drugs
* No other concurrent treatment to prevent mouth sores

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 195 (Actual)
Dates: Start 2004-04; Primary Completion 2006-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the modified Walsh mucositis scale | Length of study
  The primary aim of drug efficacy will be measured by the area under the curve (AUC) of the modified Walsh mucositis scale. Scores will be assigned for each region of oral mucosa and totaled for daily score. AUC will be obtained by graphing the total scores recorded every day during follow-up, linking time adjacent points by a straight line and calculating the area under the resulting polygon. The measurement of AUC incorporates both severity and duration of symptoms.

SECONDARY OUTCOMES:
Two sample t test and the Wilcoxon sum test. | Length of study
  Total amount of narcotics used, days of total TPN and NG feedings in patients who receive Traumeel® S and placebo will be compared. The statistical tests to be applied are the two sample t test and the Wilcoxon sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Susan F. Sencer, MD, Study Chair — Children's Hospitals and Clinics of Minnesota - Minneapolis; Indira Sahdev, MD, Study Chair — Schneider Children's Hospital
Locations (44):
- United States (37):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford Comprehensive Cancer Center at Stanford University Medical Center, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Schneider Children's Hospital, New Hyde Park, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
- Australia (3):
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Result] Sencer SF, Zhou T, Freedman LS, Ives JA, Chen Z, Wall D, Nieder ML, Grupp SA, Yu LC, Sahdev I, Jonas WB, Wallace JD, Oberbaum M. Traumeel S in preventing and treating mucositis in young patients undergoing SCT: a report of the Children's Oncology Group. Bone Marrow Transplant. 2012 Nov;47(11):1409-14. doi: 10.1038/bmt.2012.30. Epub 2012 Apr 16. PMID 22504933